CLINICAL TRIAL: NCT06630182
Title: Evaluation of the Impact of Psychological Profile on Diabetic Foot Wound Healing. Prospective, Monocentric Study
Acronym: BORTNER PIED 2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUILLET 2024
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; Foot Wound
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Foot Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 2 diabetic patients with foot wounds: Patients with type 2 diabetes referred for management of a new diabetic foot wound
  Interventions: Other: Bortner self-questionnaire; Other: Self-questionnaire BFI-10

INTERVENTIONS:
Other: Bortner self-questionnaire — 14 items
Other: Self-questionnaire BFI-10 — 10 items

SUMMARY:
Foot wounds in patients with diabetes are one of the most frequent complications associated with diabetes. Despite the progress made in its management in recent years, the risk of amputation remains high in cases of diabetic foot wounds.

Several studies have highlighted the value of analyzing the psychological profile A or B, defined by self-questionnaire using Bortner's method. The A personality profile is characterized by hyperactivity, combativeness and exaggerated ambition, while the B profile is characterized by less sensitivity to stress and reduced combativeness.

Type A personality profile is associated with reduced cardiovascular mortality in type 1 diabetes. Type B personality profiles have also been shown to be associated with inflammation in both type 1 and type 2 diabetes.

Our group showed that patients with diabetes and a foot wound were more likely to have a type B psychological profile than patients with diabetes and no foot wound.

However, to our knowledge, it has never been determined whether the psychosomatic profile type A or B assessed by the Bortner self-questionnaire influenced wound healing and the risk of amputation.

The aim of this study is to determine whether type A or B psychosomatic profile influences wound healing in diabetic feet.

This study will be carried out in the endocrinology, diabetology and nutrition department of the Dijon Bourgogne University Hospital. 308 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given his non-opposition
* Person over 18 years of age
* Person with type 2 diabetes
* Person referred for management of a new diabetic foot wound

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant women, women in labour or breastfeeding mothers
* An adult who is incapable or unable to give consent
* Minors
* Person unable to complete self-questionnaires

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with type 2 diabetes referred for management of a new diabetic foot ulcer
Sampling Method: Non-Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Bortner self-questionnaire score | At 6 months
  Comparison of the Bortner self-questionnaire score in subjects with a healed diabetic foot wound and those with an unhealed foot wound.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France